CLINICAL TRIAL: NCT06818214
Title: Mechanistic Study on the Diagnosis of Esophageal Cancer Lymph Node Metastasis Using Spectral CT, Multimodal MRI, FAPI PET-CT, Pathology, and AI Evaluation System
Status: Not yet recruiting | Type: Observational
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Qujinrong, Dr., Henan Cancer Hospital
Other Study IDs: 2024-527
Record Dates: First submitted 2025-01-21; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the group with lymph node metastasis in esophageal cancer
- the group without lymph node metastasis in esophageal cancer

SUMMARY:
The objective of this study is to address the urgent issues in the diagnosis of lymph node metastasis in esophageal cancer. By employing multimodal MRI, spectral CT imaging and FAPI PET-CTtechniques, the study will correlate lymph node images with postoperative pathology results. Additionally, AI technology will be applied to learn from multimodal imaging data, enabling comprehensive analysis and evaluation of lymph node metastasis. Using a large volume of clinical and imaging data, a predictive model will be established to provide individualized lymph node metastasis risk assessments for each esophageal cancer patient. This will, in turn, offer robust support for personalized treatment strategies in esophageal cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients with pathological diagnosis of esophageal cancer.
2. Patients underwent radical esophagectomy and lymph node dissection, with preoperative multimodal MRI, spectral CT and FAPI PET-CT ; patients underwent neoadjuvant therapy followed by radical surgery, with preoperative multimodal MRI, spectral CT and FAPI PET-CTboth before and after neoadjuvant therapy.
3. No history of malignant tumors or cancer-related treatments.
4. Complete postoperative pathological data, allowing for a one-to-one comparison of preoperative lymph node imaging and postoperative histopathology for evaluation.

Exclusion Criteria:

1. Contraindications for MRI, spectral CT or FAPI PET-CT.
2. Patients who refuse to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients are from the Esophageal Cancer Diagnosis and Treatment Center of the Affiliated Tumor Hospital of Zhengzhou University. Data will be collected from Feburary 2025 to January 2030, from patients with biopsy-confirmed esophageal cancer. Based on clinical needs, initial staging will be performed through EUS, spectral CT, or PET-CT. Patients who are planned for direct surgery will undergo MRI within 7 days prior to surgery; patients who are planned for neoadjuvant therapy will undergo spectral CT and MRI examinations both before neoadjuvant therapy and within 7 days before surgery.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2030-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
MRI, spectral CT and FAPI PET-CT combined with AI in prediction of lymph node status in esophageal cancer | February 2025 - January 2030
  To evaluate the effectiveness of multimodal MRI, spectral CT imaging, and FAPI PET-CT combined with AI in determining the preoperative lymph node status (presence or absence of metastasis) in patients with esophageal cancer, with confirmation through pathological assessment.

IPD SHARING:
Plan to Share IPD: Undecided